CLINICAL TRIAL: NCT05279196
Title: Biological Variables Associated With the Response to Intensive Training in Athletes (CareStress)
Brief Title: Biological Variables Associated With the Response to Intensive Training in Athletes
Acronym: CareStress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21_0102
Record Dates: First submitted 2022-03-03; First posted 2022-03-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Muscle Injury

STUDY DESIGN:
Intervention Model Description: Comparative study of two groups of subjects formed a posteriori from a cohort follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscular response to the training (Experimental): Epigenetic signature associated with different levels of muscle response induced by 6-month training
  Interventions: Other: Quadriceps microbiopsy and blood collection

INTERVENTIONS:
Other: Quadriceps microbiopsy and blood collection — Microbiopsy of the quadriceps muscle using a needle, "Tru-cut" biopsy, associated with a blood sampling at the start and after 6 months of a muscle strengthening training program

SUMMARY:
There is in humans, at the muscular level, a great interindividual variability in response to the same mechanical stress. This phenotypic variability is multifactorial, influenced by environmental factors as well as multiple genetic variants. Thus, for the same level of muscle damage, two subjects with the same anthropometric characteristic, the same age, with the same medical history and the same level of physical activity, will present a variable level of muscle regeneration underpinned by the biological function of muscular stem cells and their microenvironment. Thus, faced with the same training, some athletes will develop iterative muscular lesions and more disabling repair deficits than others without knowing the reason of this greater susceptibility.

Indeed, the links between the genotype of the skeletal muscle fiber and its response to exercise, as well as the regulation of muscle mass are poorly understood. Yet, in young adults, up to 70% of the observed variability in muscle strength and size is hereditary. This heritability of muscle size and strength seems to be lower in older people, probably related to increased comorbidity. Numerous experiments with athletes subjected to the same resistance exercise training have identified good and bad hypertrophic skeletal muscle responders. However, genetic variants that contribute to skeletal muscle strength and mass are largely understudied while a growing body of evidence indicates that epigenetic effectors, which modulate gene expression, may contribute to human muscle response heterogeneity to the same mechanical stress. Thus, to date, no analysis of the role of the interaction between genetic and epigenetic factors involved in the muscle functional response to exercise exists. The main hypothesis is that the epigenetic status of muscle stem cells (satellite cells) is an important contributor in muscle mass response to exercise by modulating chromatin architecture.

Thus this study will identify the epigenetic modifications induced by training and their interaction with the genetic factors involved in the response of the biological function of the satellite cells to this training and on the other hand, to be able to link it to a blood signature.

DETAILED DESCRIPTION:
The study will be carried out in close collaboration with the Director of the Expertise and Sports Performance Center (CREPS) of Montpellier. Compared to the athlete's usual seasonal training program, his participation in research will be limited to two visits to the Montpellier University Hospital where a quadriceps micro biopsy and a blood test will be carried out. During the first visit to the Montpellier University Hospital, a short clinical examination will also be carried out including an interrogation on his medical history, his consumption of drugs, alcohol, tobacco as well as the measurement of his weight and height and a simple cardiopulmonary auscultation. As part of the standard care for athletes, the training program carried out at CREPS Montpellier will be defined by weekly strength exercises to increase muscle mass. As part of this program and approximately one week before the two visits to the Montpellier University Hospital, an evaluation of the mass and the contractile function of the muscle will be carried out. The measurement of muscle mass will be carried out by Magnetic Resonance Imaging. The contractile function of the quadriceps muscle will be measured on a weight bench equipped with a dynamometer at the CREPS in Montpellier. Data from these assessments will be collected as part of the research.

This study will allow the synthesis of a muscular organoid, representative of an in vivo muscle, allowing the in vitro study of muscular lesions associated with the rupture of muscle fibres and the activation of satellite cells allowing the regeneration of damaged fibres. This in vitro muscle model will allow us to evaluate the inter-individual variability of the muscle response to the same mechanical stress and to study its link with the dynamic epigenetic changes specific to each athlete. This study will make it possible, for the first time, to evaluate whether an epigenetic signature predictive of the muscular response to an injury could also be found in blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Senior male athlete aged between 40 and 60 inclusive
* Athlete following a program over a season of muscle building at CREPS, the objective of which is to improve their performance in a middle-distance race.

Exclusion Criteria:

* Subject having a contraindication to follow the complete muscle building program at CREPS with in particular a contraindication to the measurement of muscle mass by Magnetic Resonance Imaging
* Subject presenting all criteria which can by themselves alter the function of the respiratory muscles such as chronic obstructive pulmonary disease, heart failure, systemic infection, neuromuscular pathology, psychiatric pathology, metabolic disorder.
* Subjects with coagulopathy or thrombocytopenia.
* Use of anabolic drugs to increase muscle mass
* Subject suspected of doping
* Subject allergic to xylocaine

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
DNA methylation profile of satellite cells associated with a gain in muscle mass | 6 months
  DNA methylation profile of satellite cells from the quadriceps obtained from athletes at the start and after 6 months of training, will be determine using DNA methylation profiling microarray.
  Two groups of athletes will be constituted according to the gain (in % compared to the initial value) in muscular strength of the quadriceps induced by the training and evaluated on a strength bench.
  In order to identify a DNA methylation signature associated to the gain in muscle mass, DNA methylation profile will be compared between athletes considered to be good or bad responders to training.

SECONDARY OUTCOMES:
Number and size of myoblasts obtained per satellite cells from the quadriceps | 6 months
  Satellite cells derived from quadriceps biopsy in athletes at the start and after 6 months of training will be placed in a culture dish treated with type 1 collagen in a thin layer of matrigel. After culture, proliferation and differentiation of myoblast cells will be assessed by cell counting and immunofluorescence with antibodies directed against muscle markers.
Comparison of number and size of myoblasts obtained in vitro and the muscular response to training in the same athlete | 6 months
  Size of myotubes regenerated in vitro from satellite cells taken from athletes after 6 months of training will be compared to the gain in muscle mass, strength and endurance of the quadriceps induced by training in the same athlete.
Comparison of the DNA methylation profile of satellite cells from the quadriceps and blood mononuclear cells in the same athlete | 6 months
  DNA methylation profile of satellite cells from the quadriceps and blood mononuclear cells obtained from athletes at the start and after 6 months of training, will be determine using DNA methylation profiling microarray. DNA methylation profile obtained from satellite cells and mononuclear cells in a same athlete will be compared to identify a correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No